CLINICAL TRIAL: NCT02749123
Title: Comparison of Prescription Lidocaine Patch to Over the Counter Lidocaine Patch and Placebo for Back Pain and Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: J.A.R. Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 527-03
Record Dates: First submitted 2016-04-18; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Back Pain; Arthritis
MeSH Terms: conditions — Back Pain; Arthritis | interventions — Lidocaine; Transdermal Patch; Lidoderm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine5% v Lidocaine3.6%,Menthol1.25% (Active Comparator): Daily patch Q12 followed by Q12 of no patch
  Interventions: Drug: lidocaine 5% patch; Drug: lidocaine 3.6%, menthol 1.25%
- Lidocaine 3.6%, menthol 1.25% v placebo (Placebo Comparator): Daily patch Q12 followed by Q12 of no patch
  Interventions: Drug: lidocaine 3.6%, menthol 1.25%; Drug: Placebo

INTERVENTIONS:
Drug: lidocaine 5% patch — 10cmx 14 cm transdermal patch sealed in its own pouch
  Other Names: Lidoderm
  Arms: Lidocaine5% v Lidocaine3.6%,Menthol1.25%
Drug: lidocaine 3.6%, menthol 1.25% — 10cmx 14 cm transdermal patch sealed in its own pouch
  Other Names: LidoPatch
Drug: Placebo — patch with no active manufactured to have the same look and feel as Lidoderm 10cmx 14 cm transdermal patch sealed in its own pouch
  Arms: Lidocaine 3.6%, menthol 1.25% v placebo

SUMMARY:
A comparison of transdermal patches for efficacy, side effects and quality of life for patients with back pain and arthritis. The three arms in the trial were; prescription strength lidocaine 5%, over the counter lidocaine 3.6%, menthol 1.25% and placebo.

DETAILED DESCRIPTION:
In this comparison of; lidocaine 5%, lidocaine/menthol 1.25% and placebo for patients with back pain and arthritis, subjects had to qualify by meeting various inclusion and exclusion criteria. Subjects signed an informed consent and were randomized in a double blinded fashion to one of the three arms. After randomization subjects completed a baseline questionnaire regarding how pain affects their lives. Then they began therapy with their blinded product. This same questionnaire was administered after the second day of therapy and after the final day on day 10. Responses at the day two and ten endpoints were compared to baseline to access the response of each arm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of back pain
* Diagnosis of arthritis

Exclusion Criteria:

* Pregnancy or expected pregnancy in the next three months
* Allergic to any lidocaine, menthol and methylparaben
* No reliable access to the internet
* Baseline average pain intensity of 1,2,9 or 10 on a scale of 0-to 10.
* Pain on the area of the body not conducive to patch therapy (eg fingers, toes etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy comparison of lidocaine 5% and lidocaine 3.6%, menthol 1.25% as measured by VAS numeric 0-10 pain scale | Day ten
  Endpoint is a non-inferiority statistical comparison. Comparison is based off of analysis of identical questionnaires administered at baseline and day ten

SECONDARY OUTCOMES:
Quality of life comparison of placebo and lidocaine 3.6%, menthol 1.25% as measured by VAS numeric 0-10 pain scale | Day ten
  Statistical superiority sought for lidocaine 3.6%,menthol 1.25% compared to placebo. Comparison is based off of analysis of identical questionnaires administered at baseline and day ten.
Efficacy comparison of placebo and lidocaine 3.6%, menthol 1.25% as measured by VAS numeric 0-10 pain scale | Day 10
  Statistical superiority sought for lidocaine 3.6%,menthol 1.25% compared to placebo. Comparison is based off of analysis of identical questionnaires administered at baseline and day ten.
Side effect comparison of placebo and lidocaine 3.6%, menthol 1.25% as measured by VAS numeric 0-10 pain scale | Day 10
  Endpoint is a non-inferiority statistical comparison. Comparison is based off of analysis of identical questionnaires administered at baseline and day ten.
Side effect comparison of lidocaine 5% and lidocaine 3.6%, menthol 1.25% as measured by VAS numeric 0-10 pain scale | Day 10
  Endpoint is a non-inferiority statistical comparison. Comparison is based off of analysis of identical questionnaires administered at baseline and day ten.

CONTACTS AND LOCATIONS:
Locations (1):
- Advocate Good Sheppard Hospital, Barrington, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Investigators plan to share the study results as a whole but no plans to share individual results.